CLINICAL TRIAL: NCT06220955
Title: Quantification of the Differences in the Diagnostic Relationships Between Centric Occlusion Versus Maximum Intercuspation in Adult Orthodontic Patients : A Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Elzanaty, resident, Cairo University
Other Study IDs: ORTH 7-1-1
Record Dates: First submitted 2023-12-08; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Centric Relation Registration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: centric relation registration — centric relation registration using conventional and digital methods
Other: maximum intercuspation registration — maximum intercuspation registration

SUMMARY:
The aim of the study is to quantify the differences in the diagnostic relationships between Centric occlusion versus maximum intercuspation in adult orthodontic patients with Cetric relation recoded using both conventional method utilizing semi-adjustable articulator and face bow record in addition to digital method proposed by Radu et al for finding and recording CR using a dental intraoral scanner with a leaf gauge

DETAILED DESCRIPTION:
Study design Cross-sectional study PICO Components P: Adult orthodontic patient I: Centric occlusion C: Maximum intercuspation

O: -orthodontic relations:

Molar relation Canine relation Incisor relation Overjet Overbite Midline discrepancy

ELIGIBILITY:
Inclusion Criteria:

orthodontic patient having full permanent dentition

Exclusion Criteria:

* patients who had undergone previous orthodontic treatment, and syndromic patients, retained primary teeth , teeth heavily restored

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: rthodontic patient having full permanent dentition
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
overjet | 1 day between the maximum intercuspation and centric relation records
  overjet change measurement in millimeter

SECONDARY OUTCOMES:
overbite | 1 day between the maximum intercuspation and centric relation records records
  measurement in millimeter
midline shift | 1 day between the 2 records
  superimposition of both centric relation and maximum intercuspation digitally
incisor relation | 1 day between the maximum intercuspation and centric relation records records
  measurement in millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No